CLINICAL TRIAL: NCT05698836
Title: Cardiovascular Health Assessment of Preterm- and TERm-born Children
Acronym: CHAPTER
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 18/WM/0131
Record Dates: First submitted 2022-10-31; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-10

CONDITIONS: Premature Birth
Keywords: cardiac function; preterm; children
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the CHAPTER study is to help understand how complications during pregnancy, such as preterm birth, affect how childrens' hearts and blood vessels develop.

DETAILED DESCRIPTION:
Young adults born preterm (less than 37 weeks gestation) have alterations in the structure and function of the heart, with similar changes observed in preterm infants in the first three months of life. It is unknown whether these early changes in the heart seen in the first few months of life are relevant to long-term changes in heart structure and function. Heart changes have also not been well studied in children born preterm. To investigate this, the study will follow up children from the EPOCH study and will perform two study visits for each child (n=100 preterm and n=100 term) that will use echocardiography and cardiovascular magnetic resonance. Individuals in the EPOCH study had echocardiography measures done at birth and three months postnatal age. It will therefore be possible to do longitudinal echocardiography measures from birth up to ages 12 years to determine whether postnatal heart changes in preterm infants track into childhood. Cardiovascular magnetic resonance will allow for the determination of whether these early heart changes influence heart pump function. Finally, by measuring lung function, blood vessel structure and function, and blood pressure, it will be possible to determine how heart changes relate to other components of the cardiovascular system. This data will be used to confirm the relevance of early heart remodelling in preterm-born offspring over time and provide more comprehensive heart phenotyping for preterm-born children. Together, this information can be used to design future intervention strategies in preterm-born individuals to reduce cardiovascular risk in this growing subgroup of the population.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent or legal guardian gives consent and the participant, where age-appropriate, gives assent for participation in the study.
* Participant is male or female, aged 3-9 years at enrolment.
* Participant previously took part in the EPOCH study, or the participant's friend or sibling took part.

Exclusion Criteria:

* Evidence of congenital heart disease or significant chronic disease relevant to cardiovascular or metabolic status

For exclusion of MRI component only:

* Contraindication to MRI
* Unsuitable for MRI based on the responses to the MRI screening form

Ages: 3 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Children aged 3--12 years old born preterm (less than 37 weeks gestation) or term (37--42 weeks gestation) delivered at or admitted to the Oxford University Hospitals NHS Foundation Trust who took part in the EPOCH study. Recruitment also includes both siblings and friends of those who took part in the original EPOCH study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2036-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac left ventricular mass | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of left ventricular mass indexed to body surface area (in g and g/m^2)

SECONDARY OUTCOMES:
Cardiac right ventricular mass | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of right ventricular mass indexed to body surface area (in g and g/m^2)
Cardiac left ventricular end-diastolic volume | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of cardiac left ventricular end-diastolic volume indexed to body surface area (in ml and ml/m^2)
Cardiac right ventricular end-diastolic volume | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of cardiac right ventricular end-diastolic volume indexed to body surface area (in ml and ml/m^2)
Cardiac left ventricular systolic function | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of left ventricular systolic function: left ventricular ejection fraction (in %)
Cardiac right ventricular systolic function | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of right ventricular systolic function: tricuspid annular plane systolic excursion (in cm)
Cardiac left ventricular diastolic function | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of right ventricular (RV) diastolic function: RV Doppler early/late diastolic tricuspid inflow velocity ratio (E/A)
Cardiac right ventricular diastolic function | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Echocardiography assessment of left ventricular (LV) diastolic function: LV Doppler early/late diastolic mitral inflow
Morphology of the left ventricles | 6-9 years of age
  MRI assessment of the left ventricles morphology using cardiac statistical atlas and principal component analysis
Morphology of the right ventricles | 6-9 years of age
  MRI assessment of the right ventricles morphology using cardiac statistical atlas and principal component analysis
Cardiac flow dynamics of the left ventricle | 6-9 years of age
  MRI assessment of direct flow, delayed ejection flow, retained inflow, residual volume kinetic energy flow components at end diastole (measured at end diastole in mJ and overall % contribution)
Systolic blood pressure measurement | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Resting brachial blood pressure measurement (in mmHg)
Diastolic blood pressure measurement | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Resting brachial blood pressure measurement (in mmHg)
Mean arterial pressure | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  The average arterial pressure from resting brachial blood pressure measurement (in mmHg)
Retinal arteriolar structure | 6-9 years of age
  Central retinal arteriolar equivalent (CRAE in μm) measured using retinal imaging
Retinal venular structure | 6-9 years of age
  Central retinal venular equivalent (CRVE in μm) measured using retinal imaging
Retinal arteriolar-to-venular diameter ratio (AVR) | 6-9 years of age
  The ratio of average retinal arteriolar diameter (CRAE in μm) and average retinal venous diameter (CRVE in μm) measured using retinal imaging
Lung function | 6-9 years of age
  The forced expiratory volume in one second (FEV1 in L), forced vital capacity (FVC in L), and the ratio of FEV1 to FVC (FEV1/FVC) measured using spirometry
Objective measure of physical activity | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  The amount of moderate to vigorous physical activity (in h/week) and vigorous physical activity (in h/week) measured using wrist worn accelerometer
Body weight | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Body weight measured in kg
Body height | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Body weight measured in m
Body mass index | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Body weight divided by the square of height (in kg/m2)
Mid-arm circumference | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  Mid-arm circumference measured in cm
Waist-to-hip ratio | 3-5 years of age OR 8-12 years of age; AND 6-9 years of age
  The ratio of waist circumference (in cm) to hip circumference (in cm)

OTHER OUTCOMES:
Tube formation capacity in endothelial colony forming cells (ECFCs) | 6-9 years of age
  The number of closed tubes formed/1.5x10^4 cells
Endothelial colony forming cells (ECFC) branches formed | 6-9 years of age
  The number of branches formed/1.5x10^4 cells
Endothelial colony forming cells (ECFC) colony formation | 6-9 years of age
  Days for ECFC colony formation, measured in days
Endothelial colony forming cells (ECFC) proliferation rate | 6-9 years of age
  ECFC proliferation rate, measured as a percentage
Subcortical brain volume of hippocampus | 6-9 years of age
  Subcortical brain volume of hippocampus (in mm3) assessed on T1-weighted sequence of brain MRI
Subcortical brain volume of thalamus | 6-9 years of age
  Subcortical brain volume of thalamus (in mm3) assessed on T1-weighted sequence of brain MRI
White matter hyperintensities count | 6-9 years of age
  The number of white matter hyperintensities on T2-weighted sequence of brain MRI
White matter hyperintensities volume | 6-9 years of age
  Total volume of white matter hyperintensities (in mm3) assessed on T2-weighted sequence of brain MRI
Cerebral vessel lumen diameter | 6-9 years of age
  Cerebral vessel lumen diameter (in μm) assessed on the time-of-flight sequence of brain MRI
Cerebral vessel density | 6-9 years of age
  Cerebral vessel density (in mm3) assessed on the time-of-flight sequence of brain MRI
Cerebral vessel tortuosity | 6-9 years of age
  The ratio of cerebral vessel tortuosity assessed on the time-of-flight sequence of brain MRI
Whole brain grey matter perfusion or cerebral blood flow (CBF) | 6-9 years of age
  Whole brain grey matter perfusion/CBF (in ml/100g/min) assessed on arterial spin labelling of brain MRI
Arterial cerebral blood volume fraction | 6-9 years of age
  Arterial cerebral blood volume fraction (in %) assessed on arterial spin labelling of brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lewandowski, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No